CLINICAL TRIAL: NCT02518516
Title: Use of High Potency Statins and Rates of Admission for Acute Kidney Injury: Multicenter, Retrospective Observational Analysis of Administrative Databases
Brief Title: High Potency Statins and Acute Kidney Injury
Status: Completed | Type: Observational
Sponsor: Canadian Network for Observational Drug Effect Studies, CNODES (Other)
Collaborators: Drug Safety and Effectiveness Network, Canada (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: CNODES_Demo_1
Record Dates: First submitted 2015-08-04; First posted 2015-08-07 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2015-08

CONDITIONS: Hypercholesterolemia
Keywords: Statins, HMG-CoA; Acute kidney injury; Kidney diseases; Renal failure
MeSH Terms: conditions — Hypercholesterolemia; Acute Kidney Injury; Kidney Diseases; Renal Insufficiency | interventions — Rosuvastatin Calcium; Atorvastatin; Simvastatin; Fluvastatin; Pravastatin; Lovastatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- High potency statin users: Exposure will be defined as a new prescription for a high dose statin (rosuvastatin, high doses of atorvastatin, and high doses of simvastatin between 1 January 1997 and 30 of April 2008, or 1 year after the beginning of data availability.
  Interventions: Drug: Rosuvastatin (≥10 mg); Drug: Atorvastatin (≥20 mg); Drug: Simvastatin (≥40 mg)
- Low potency statin users: Exposure will be defined as a new prescription for a low dose statin (all doses of fluvastatin, all doses of pravastatin, all doses of lovastatin; low doses of atorvastatin and simvastatin) between 1 January 1997 and 30 of April 2008, or 1 year after the beginning of data availability.
  Interventions: Drug: Fluvastatin; Drug: Pravastatin; Drug: Lovastatin; Drug: Atorvastatin (<20mg); Drug: Simvastatin (<40 mg)

INTERVENTIONS:
Drug: Rosuvastatin (≥10 mg) — Current cumulative exposure to high dose rosuvastatin (ATC C10AA07) will be defined as a prescription for ≥10 mg of rosuvastatin dispensed prior to the index date in one of the following exposure duration categories (≤120 days, 121-365 days, or 366-730 days).
  Past exposure to high dose rosuvastatin (ATC C10AA07) will be defined as a prescription for ≥10 mg of rosuvastatin dispensed >120 days of the index date (i.e. no exposure within 120 days of the index date).
  Groups: High potency statin users
Drug: Atorvastatin (≥20 mg) — Current cumulative exposure to high dose atorvastatin (ATC C10AA05) will be defined as a prescription for ≥20 mg of atorvastatin dispensed prior to the index date in one of the following exposure duration categories (≤120 days, 121-365 days, or 366-730 days).
  Past exposure to high dose atorvastatin (ATC C10AA05) will be defined as a prescription for ≥20 mg of atorvastatin dispensed >120 days prior to the index date (i.e. no exposure within 120 days of the index date).
  Groups: High potency statin users
Drug: Simvastatin (≥40 mg) — Current cumulative exposure to high dose simvastatin (ATC C10AA01) will be defined as a prescription for ≥40 mg simvastatin dispensed prior to the index date in one of the following exposure duration categories (≤120 days, 121-365 days, or 366-730 days).
  Past exposure to high dose simvastatin (ATC C10AA01) will be defined as a prescription for ≥40 mg simvastatin dispensed >120 days prior to the index date (i.e. no exposure within 120 days of the index date).
  Groups: High potency statin users
Drug: Fluvastatin — Current cumulative exposure to fluvastatin (ATC C10AA04) will be defined as a prescription for any dose of fluvastatin dispensed prior to the index date in one of the following exposure duration categories (≤120 days, 121-365 days, or 366-730 days).
  Past exposure to fluvastatin (ATC C10AA04) will be defined as a prescription for any dose of fluvastatin dispensed >120 days prior to the index date (i.e. no exposure within 120 days of the index date).
  Groups: Low potency statin users
Drug: Pravastatin — Current cumulative exposure to pravastatin (ATC C10AA03) will be defined as a prescription for any dose of pravastatin dispensed prior to the index date in one of the following exposure duration categories (≤120 days, 121-365 days, or 366-730 days).
  Past exposure to pravastatin will be defined as a prescription for any dose of pravastatin (ATC C10AA03) dispensed >120 days prior to the index date (i.e. no exposure within 120 days of the index date).
  Groups: Low potency statin users
Drug: Lovastatin — Current cumulative exposure to lovastatin (ATC C10AA02) will be defined as a prescription for any dose of lovastatin dispensed prior to the index date in one of the following exposure duration categories (≤120 days, 121-365 days, or 366-730 days).
  Past exposure to lovastatin will be defined as a prescription for any dose of lovastatin (ATC C10AA02) dispensed >120 days prior to the index date (i.e. no exposure within 120 days of the index date).
  Groups: Low potency statin users
Drug: Atorvastatin (<20mg) — Current cumulative exposure to low dose atorvastatin (ATC C10AA05) will be defined as a prescription for <20 mg of atorvastatin dispensed prior to the index date in one of the following exposure duration categories (≤120 days, 121-365 days, or 366-730 days).
  Past exposure to low dose atorvastatin (ATC C10AA05) will be defined as a prescription for <20 mg of atorvastatin dispensed >120 days prior to the index date (i.e. no exposure within 120 days of the index date).
  Groups: Low potency statin users
Drug: Simvastatin (<40 mg) — Current cumulative exposure to low dose simvastatin (ATC C10AA01) will be defined as a prescription for <40 mg simvastatin dispensed prior to the index date in one of the following exposure duration categories (≤120 days, 121-365 days, or 366-730 days).
  Past exposure to low dose simvastatin (ATC C10AA01) will be defined as a prescription for <40 mg simvastatin dispensed >120 days prior to the index date (i.e. no exposure within 120 days of the index date).
  Groups: Low potency statin users

SUMMARY:
Statins are a class of cholesterol lowering medications that are prescribed for the prevention and treatment of cardiovascular disease. The purpose of this study is to determine if there is an excess risk of acute kidney injury (AKI) with high potency statins compared to low potency statins.

The investigators will carry out separate population based cohort studies using administrative health care databases in nine jurisdictions in Canada, the US, and the UK. Cohorts will be defined by the initiation of a statin, with follow-up until hospitalization for AKI. Analyses will be done separately for groups of patients with and without chronic kidney disease. The results from the separate sites will be combined in a meta-analysis to provide an overall assessment of the risk of AKI in new statin users.

DETAILED DESCRIPTION:
The study objective is to determine whether the use of high potency statins, compared with the use of low potency statins, is associated with an increased risk of acute kidney injury (AKI) in routine clinical practice. The investigators will use a common-protocol approach to conduct retrospective cohort studies using health care data from nine jurisdictions (the Canadian provinces of Alberta, British Columbia, Manitoba, Nova Scotia, Ontario, Quebec, and Saskatchewan, as well as the United States (US) MarketScan and the United Kingdom (UK) Clinical Practice Research Datalink [CPRD]). The Canadian provincial databases contain information on physician billing, diagnoses and procedures from hospital discharge abstracts, and dispensations for prescription drugs at a population level. The CPRD is a clinical database that is representative of the UK population and contains the records for patients seen at over 680 general practitioner practices in the UK; these data will be linked to the Hospital Episode Statistics (HES) database, which contains in-hospital diagnosis and procedure data.

Study population

In each jurisdiction, the investigators will assemble a study cohort that includes all patients with a new prescription for a statin, including simvastatin, lovastatin, pravastatin, fluvastatin, atorvastatin, and rosuvastatin, from the earliest availability of data at each site to the last date of available data. The date of study cohort entry is defined by the prescription date of the newly-prescribed statin.

For the purpose of this study, two separate cohorts will be created based on the presence or absence of a history of chronic kidney disease at any time prior to and including the date of study cohort entry. Chronic kidney disease is defined as patients who have 1 hospitalization or 1 physician claim 3 years prior to study cohort entry with any of the following diagnoses and corresponding diagnostic codes: chronic or unspecified renal failure (ICD-9: 585, 586; ICD-10: N18, N19), hypertensive renal disease (ICD-9: 403.x1, 404.x2, 404.x3; ICD-10: I12.0, I13.1), nephritis and nephropathy (ICD-9: 582, 583; ICD-10: N03, N05), renal sclerosis or disorder from impaired renal function (ICD-9: 587, 588; ICD-10: S00-T98). Patients in each cohort will be followed from the date of study cohort entry until an event (defined below) or censoring due to death, departure from the database, 24 months after initiation of statin treatment, a dispensing for cerivastatin, or the end of the study period (31 March 2010 or the last date of data availability at that site), whichever occurs first. Data from Alberta, Ontario, and Nova Scotia will be restricted to patients aged 65 years and older as prescription data are not available for younger patients.

Case-control selection

The cohorts defined above will be analyzed using a nested case-control analysis, where cases are defined as a hospitalization for AKI. Risk set sampling will be used to randomly select up to 10 controls for each case, matched on sex, age (± one year; however, if no controls are available, within five years), cohort entry (± 90 days), and duration of follow-up.

Exposure assessment

The exposure categories will be separated by statin potency (high vs. low dose), and the duration of current and past exposure. For all cases and controls, exposure will be defined hierarchically; more specifically, patients who receive both a high and low potency statin within the same exposure category will be classified as high potency statin users. Current use of a high potency statin will be defined by the last prescription for a high dose statin within the 60 days prior to the index date.

Current users will be further classified into three mutually exclusive durations of current exposure (≤120, 121-365, and 366-730 days). Past exposure will be defined as a new prescription for a statin at least 120 days prior to the index date.

Statistical analyses

All analyses will be conducted separately among patients with and without a history of chronic kidney disease. Conditional logistic regression will be used to estimate the odds ratios and corresponding 95% confidence intervals (CIs) of the association of hospitalization for AKI, comparing current and past use of high potency statins to low potency statins. This is considered the primary analysis. Several sensitivity analyses will be performed to assess the robustness of study results and address some of the study limitations.

High dimensional propensity scores will be estimated for all patients in the cohorts using logistic regression. Fixed cohort analyses will also be conducted on the cohorts in each jurisdiction, where the statin exposure category will be defined by the initial prescription at cohort entry. Finally, all site-specific estimates will be meta-analyzed using fixed or random-effects models with inverse variance weighting. The amount of between-site heterogeneity will be estimated using the I square statistic.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a new prescription for a statin from the earliest availability of data at each site to the last date of availability of data +365 days
* Patients who are at least 40 years of age at cohort entry
* Patients with at least one year of history in the database

Exclusion Criteria:

* Patients under the age of 40 (<66 in jurisdictions with drug data for seniors only)
* Patients with less than one year of history in the database
* Patients who received any cholesterol lowering drugs (including fibrates, niacin and ezetimibe) or underwent dialysis or a kidney transplant in the previous year

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In each jurisdiction, the investigators will assemble a study cohort that includes all patients with a new prescription for a statin, including simvastatin, lovastatin, pravastatin, fluvastatin, atorvastatin, and rosuvastatin between 1 January 1997 (or one year after the beginning of data availability) and 30 April 2008. The date of study cohort entry is defined by the prescription date of the newly-prescribed statin. Two separate cohorts will be created based on the presence or absence of a history of chronic kidney disease.
Sampling Method: Probability Sample
Enrollment: 2067639 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Number of patients hospitalized for acute kidney injury | Patients will be followed from the date of study cohort entry until either hospitalization for acute kidney injury or censoring (whichever occurs first), or will be assessed for up to 24 months.
  Patients hospitalized for acute kidney injury (including but not limited to hypertensive renal disease with renal failure, chronic glomerulonephiritis, and renal sclerosis) with any of the following diagnostic codes: ICD-9 584, 584.5, 584.6, 584.7, 584.8, or 584.9; ICD-10 N17, N17.0, N17.1, N17.2, N17.8, or N17.9.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Dormuth, M.Sc., Sc.D., Principal Investigator — Departments of Anesthesiology, Pharmacology and Therapeutics, University of British Columbia, Vancouver,BC
Locations (1):
- Dept. of Anesthesiology, Pharmacology & Therapeutics (APT), University of British Columbia, Vancouver, British Columbia, Canada

REFERENCES:
- [Result] Dormuth CR, Hemmelgarn BR, Paterson JM, James MT, Teare GF, Raymond CB, Lafrance JP, Levy A, Garg AX, Ernst P; Canadian Network for Observational Drug Effect Studies. Use of high potency statins and rates of admission for acute kidney injury: multicenter, retrospective observational analysis of administrative databases. BMJ. 2013 Mar 18;346:f880. doi: 10.1136/bmj.f880. PMID 23511950
- See also: This organization's website describing general functions, other CNODES projects, and investigator profiles. — http://www.cnodes.ca